CLINICAL TRIAL: NCT00809120
Title: Investigation of Clinical Tolerance, Cardio-respiratory Response and Muscle Fatigue During Electrostimulation
Brief Title: Tolerance to Electrostimulation in COPD Patients
Acronym: TOES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Dr François Maltais, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CER20357
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2008-09

CONDITIONS: COPD
Keywords: Electrostimulation; COPD; Tolerance; Muscle fatigue; Cardio-respiratory response
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Neuromuscular Electrical stimulator (Cefar rehab 4 pro) — 50Hz 30 min 7 sessions
  Other Names: NMES

SUMMARY:
The study was designed to test the following hypothesis

Patients with high cardio-respiratory response to electrostimulation (ES), high perception of pain during ES and high ES-induced muscle fatigue, have low tolerance to ES (more difficulties to increase intensity during training).

DETAILED DESCRIPTION:
Background: Muscle electrostimulation (ES) appears as a promising alternative to general physical reconditioning in advanced COPD and its feasibility has been confirmed in this population. However, patients are not equal in tolerance to ES. Certain patients are not able to increase ES intensity during training, limiting its benefits. Furthermore, little is known about the effect of one ES training session on cardio-respiratory response, muscle fatigue and systemic inflammation in COPD patients.

Objective: To evaluate the tolerance to ES in COPD patients and to identify the physiological parameters involved in ES tolerance.

Method: We propose to conduct a prospective study including 21 COPD patients of different pulmonary severity (7 in each group of GOLD II, III and IV). Patients will be evaluated 3 times: at day 1, day 2 and day 9. In the first session, patients will be initiated to ES and evaluated in walking distance. In the second session, patients will become autonomous with ES and they will be evaluated in muscle strength and body composition. In the third session, cardio-respiratory measurements will be performed during ES and patients will be evaluated in muscle strength and systemic inflammation (blood sampling) before and after ES. Between the 2d and the 3d sessions, patients will have to perform 5 ES sessions at home (from day 3 to day 8). Tolerance (symptoms assessed with visual analogical scale (VAS)) and intensity of ES will be measured during each ES session.

Planning analysis: The main outcome will be the change in ES intensity between session 2 and 3 (delta intensity). The other end-points will be minute ventilation, heart rate, VO2 and SaO2 during ES, but also change in ES tolerance (VAS) during ES at equal ES intensity, leg muscle fatigue after ES, body composition and changes in plasmatic proteins after ES. Simple and multiple regressions analysis will be done between delta intensity and 1/cardio-respiratory response during ES, 2/muscle fatigue after ES, 3/body composition, 4/perception of pain at session 2 (VAS), 5/changes in plasmatic proteins after ES.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with COPD.
* 40 years-old and older
* Currently or previously smoking with a smoking history of at least 10 pack-years
* Subject understands and is able to read and write French or English

Exclusion Criteria:

* absence of neuromuscular pathology
* absence of vascular pathology
* absence of dermatosis on legs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Tolerance to ES = Change in ES intensity between session 2 and 3 (delta intensity) | 1 week

SECONDARY OUTCOMES:
Cardiorespiratory response during ES | 1 week
Muscle fatigue after ES | 1 week
Body composition | 1 week
Perception of pain at session 2 (symptoms on Visual Analogic Scale) | 1 week
Plasmatic proteins after ES | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Vivodtzev I, Rivard B, Gagnon P, Mainguy V, Dube A, Belanger M, Jean B, Maltais F. Tolerance and physiological correlates of neuromuscular electrical stimulation in COPD: a pilot study. PLoS One. 2014 May 9;9(5):e94850. doi: 10.1371/journal.pone.0094850. eCollection 2014. PMID 24817528